CLINICAL TRIAL: NCT05460780
Title: First-in-human Study of MATTISSE® Tissue Engineering Chamber in Adult Female After Total Mastectomy for Breast Cancer in Immediate or Delayed 2-stage Tissue Expander Reconstruction or Conversion from Implant-based to Autologous Reconstruction
Brief Title: First-in-human, Study of MATTISSE® Tissue Engineering Chamber in Adult Female Patients Undergoing Breast Reconstruction After Mastectomy for Cancer
Acronym: TIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Medical (Industry)
Collaborators: Lattice Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3121_MATFIH22
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female; Breast Cancer Prevent; Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MATTISSE TEC (Experimental): Patient included receive MATTISSE TEC
  Interventions: Device: MATTISSE TEC

INTERVENTIONS:
Device: MATTISSE TEC — Tissue engineering chamber MATTISSE

SUMMARY:
This study is a first in human, two-stage single arm non-comparative study of safety and performance.

The aim of the study is to asses the safety and the clinical performance of a new device : the MATTISSE tissu engineering chamber.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to pathology:

* Female patient over 18 Years old
* Patient who required autologous breast reconstruction:

  * Immediate unilateral reconstruction after total mastectomy for early-stage breast cancer
  * Breast reconstruction after unilateral preventive total mastectomy
  * or delayed unilateral reconstruction after total mastectomy for early-stage breast cancer with a tissue expander implantation
  * or conversion from implant-based to autologous reconstruction: Patient who had a breast implant during a previous reconstruction after total mastectomy for cancer, and who needs to change it.
* For patient with active cancer: Patient with early-stage cancer (stage 0, I or II, with tumor size < 50mm, without lymph-node involvement) needing oncological management that does not required radiotherapy after surgery on the breast area or on the flap donor site
* Patient who required Nipple sparing (NSM) or Skin sparing mastectomy (SSM) with a unique surgical approach (same for mastectomy and implant) insertion; or implant removal for patient undergoing autologous conversion, or expender removal for patient undergoing differed reconstruction.
* Autologous reconstruction using Lateral Intercostal Perforator (LICAP) flap or an intercostal thoracic artery perforation flap (LTAP) if oncological conditions do not allow for LICAP harvesting.
* Patient medically fit for surgery without significant comorbidities
* Breast cup-size less than D
* Body mass index >20 kg/m2 or patient for whom sufficient flap volume is expected according to surgeon's assessment
* Adequate hematopoietic functions

Criteria related to population:

* Subjects who have given free, informed and written consent to participate in the study;
* Patient able to answer questionnaires, able to communicate in the language of the study country;
* Subjects affiliated to a social security schema or entitled to a social security scheme.

Non-inclusion Criteria:

Pathology related criteria:

* Patient undergoing bilateral reconstruction
* Patient undergoing bilateral preventive mastectomy
* Patient undergoing simultaneous contralateral breast reduction, mastopexy, and augmentation
* Previous history of radiotherapy on the breast area or on the flap donor site
* Previous history of breast or axillary surgery that does not allow fat flap dissection
* Presence of pacemaker or metallic prosthesis making patient unsuitable for MRI
* Body mass index >30 kg/m2
* Taking medication for weight loss at the time of inclusion visit
* Presence of major medical conditions that may compromise patient's health and healing
* Diabetes and a history of gestational diabetes
* Active smoking
* Microangiopathy, Vascular history and all systemic disease (systemic Raynaud's disease)
* Patient with intertrigo or infection or alteration of the surgical site confirmed pre-operatively by clinical examination
* Allergy to anesthetics or contrast media
* Immunocompromised patient (HIV) or patient used immunosuppressants

Population related criteria

* Pregnant patient
* or breastfeeding patient or woman who has nursed a child three months within inclusion
* Participation in a clinical trial in the 3 months prior to the initial visit
* Predicted unavailability during study.
* Patient deprived of liberty or under guardianship.
* Patient unable to give consent

Medical device related criteria

* Allergy to any of the components of the medical device.

EXCLUSION CRITERIA

* Positive or suspicious extemporaneous sentinel node biopsy
* Non integrity of LICAP and LTAP vessels, showed by the pre-operative doppler
* Patient not yet implanted with MATTISSE®, whose cancer stage will finally require radiotherapy treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety objective: To assess the 6 months surgical complications rate of MATTISSE® TEC implant-based immediate breast reconstruction. Adverse events will be recorded. | 6 months post-surgery
  Minor complications include:
  * Superficial skin necrosis that requires only debridement
  * Flap necrosis
  * Subcutaneous hematoma: any hematoma requiring surgical exploration
  * Inflammatory reaction
  * Seroma: defined as that which requires echo-guided puncture at least once after drain removal.
  * Pain
  * Delayed wound healing/wound dehiscence: any wound healing problems, detected during clinical examination and not requiring an intervention
  * Implant malposition
  * Superficial Venous Thrombosis (Mondor disease)
  * Capsular contracture
  Major complications include:
  * All complications that lead to MATTISSE® TEC removal:
  * Skin necrosis leading to implant exposure
  * Infection
  * Implant malposition leading to implant exposure
  * Device failure or defect: when the implant breaks or collapses, e.g., the base separates from the shell, failure at the time of surgical placement (fracture of the TEC before placement)
  * Granuloma.
Performance objective: To assess the efficacy at 6 months post-operation of breast reconstruction using MATTISSE® breast implants in patients undergoing breast reconstitution after total mastectomy surgery for cancer. | 6 months post-surgery
  Success is defined as:
  * Tissue expansion (flap enlargement) from implantation up to 6 months post operation --> A 50% increase in the expanded size at 6 months compared to initial size flap is considered as a success. Indeed, the optimal growth of the flap is expected at 6 months,
  * Tissue expansion will be assessed using MRI at discharge (after surgery) and 6 months post operative. The volume of flap at 6 months will be compared to the flap size initially implanted. All MRI imaging will be assessed by and independent expert radiologist.
  Failure is defined as:
  * less than 50% increase in the expanded size at 6 months compared to initial size flap MATTISSE® Prothesis removal

SECONDARY OUTCOMES:
Evolution of tissue expansion (flap enlargement) from implantation up to 36 months post operation. | Surgery visit, 3, 6, 12, 24 and 36 months post-intervention
  Tissue expansion will be assessed using MRI at discharge (after surgery), 12, 24 and 36 months post operative.
  All MRI imaging will be assessed by and independent expert radiologist.
Evolution of breast softness from inclusion to 36 months | Surgery visit, 3, 6, 12, 24 and 36 months post-intervention
  * The breast softness will be assessed by investigator surgeon and patients themselves at discharge (after surgery), 3, 6 ,12, 24 and 36 months as:
  * Stage 1: Breast is soft
  * Stage 2: Breast is hard
  * Stage 3: Breast is hard with distortion
  * Stage 4: Breast is hard, painful with distortion
Evolution of MATTISSE® TEC resorption until 36 months follow up: the resorption is active between 6 and 12 months after surgery. | Surgery visit, 3, 6, 12, 24 and 36 months post-intervention
  MATTISSE® TEC resorption will be observed quantitatively on MRI achieved at 3, 6, 12, 24 and 36 months associated with the touch of the surgeon and patients feeling. The TEC resorption will be classified as:
  * Absent: no resorption at all.
  * Small resorption: TEC has been reabsorbed a little bit compared to the initial
  * Great resorption: TEC has been absorbed a lot but not totally
  * Total: Shell and base are no longer visible on the MRI and not felt by the surgeon
The volume of the reconstructed breast compared to the volume of the contralateral one at 12, 24 and 36 months | 3, 6, 12, 24 and 36 months post surgery
  At 12, 24 and 36 months, we will assess during physical examinations, the volume of the reconstructed breast and the volume of the contralateral one.
Aesthetic breast appearance before and after surgery using photo | 3, 6, 12, 24 and 36 months post surgery
  Aesthetic breast appearance will be assessed before surgery, 6 at 12, 24 and 36 months post-surgery using standardized photographs. The assessment will be done by the surgeon and 2 independent external specialists who validated standardized photographs.
  The following scoring points will be used:
  * Excellent: Treated breast nearly identical to that before surgery
  * Good: Treated breast slightly different to that before surgery
  * Fair: Treated breast clearly different to that before surgery but not seriously distorted
  * Poor: Treated breast seriously distorted compared to that before surgery
The maintain of breast (i.e., flap) volume stability at 12, 24 and 36 months compared to that at 6 months | 3, 6, 12, 24 and 36 months post surgery
  Flap volume at 12, 24 and 36 months is compared at that assessed at 6 months using MRI.
  All MRI imaging will be assessed by and independent expert radiologist.
The impact of the flap transfer on the donor site assessed at surgery, 3, 6, 12, 24 and 36months post-surgery | 3, 6, 12, 24 and 36 months post surgery
  Impact of the flap transfer on the donor site will be assessed at surgery, 3, 6, 12, 24 and 36 months post-surgery using different parameters:
  * Tissue necrosis (Yes/ No)
  * Symmetry of the donor site area (comparing to the other side of the patient): Yes/ No
Pain (VAS) | 3, 6, 12, 24 and 36 months post surgery
  Pain score will be assessed at inclusion, discharge, 3, 6, 12, 24 and 36 month using a 10 Visual Analogue Scale [VAS, 0 (no pain) and 10 (worst possible pain)]
The quality of life and the satisfaction of patients | 3, 6, 12, 24 and 36 months post surgery
  Quality of life and patients' satisfaction will be done through the BREAST-Q© questionnaire (module of reconstruction pre and post-surgery version) at inclusion and at 3, 6 and 12 months post operative. The quality of life is evaluated through 2 scales (psychological well-being and physical well-being: breast).
  The satisfaction is evaluated with 1 scale : (satisfaction with breast).
Surgeon satisfaction regarding the use of MATTISSE® TEC and implantation procedure. | Visit 2, surgery
  - Surgeons' satisfaction regarding the use of MATTISSE® TEC and implantation procedure will be assessed on: Global satisfaction of the surgeon (5 points Likert scale)
  * Ease of use
  * Material ergonomics
  * Ease of insertion
  * Ease of fixing
Evolution of biological parameters up to 6 months after surgery | Inclusion, Discharge, 3, 6 months post-intervention
  Complete blood counts evolution will be assessed at inclusion, at discharge, and at 3 and 6 months post-implantation, by measuring Hemoglobin , leukocytes Lymphocyte rate Neutrophil rate and Thrombocytes
  Units:
  * Hemoglobin : g/L
  * leukocytes :10⁹/L
  * Lymphocyte rate : %
  * Neutrophil rate : %
  * Thrombocytes : 10⁹/L
Evolution of biological parameters up to 6 months after surgery | Inclusion, Discharge, 3, 6 months post-intervention
  C-reactive protein evolution will be assessed at inclusion, at discharge, and at 3 and 6 months post-implantation, by measuring CRP
  Unit:
  - CRP : nmoL/L
Evolution of biological parameters up to 6 months after surgery | Inclusion, Discharge, 3, 6 months post-intervention
  Total protein evolution will be assessed at inclusion, at discharge, and at 3 and 6 months post-implantation, by total protein assay
  Unit:
  Total protein: Normal or Not normal
Evolution of biological parameters up to 6 months after surgery | Inclusion, Discharge, 3, 6 months post-intervention
  Protein electrophoresis will be assessed at inclusion, at discharge, and at 3 and 6 months post-implantation, by performing protein electrophoresis.
  Unit :
  Protein electrophoresis: Normal or Not normal
Safety up to 36 months post operation | Surgery visit, 3, 6, 12, 24 and 36 months post-intervention
  Safety up to 36 months, will be assessed by measuring the complication rate after breast reconstruction using MATTISSE® TEC. Adverse events up to 36 months post operation will be recorded.

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - CHU de Strasbourg, Strasbourg, France
  - Hospital of Lille, Lille, Nord
- Institute of Clinical Oncology, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harbeck N, Penault-Llorca F, Cortes J, Gnant M, Houssami N, Poortmans P, Ruddy K, Tsang J, Cardoso F. Breast cancer. Nat Rev Dis Primers. 2019 Sep 23;5(1):66. doi: 10.1038/s41572-019-0111-2. PMID 31548545
- [Background] Schmauss D, Machens HG, Harder Y. Breast Reconstruction after Mastectomy. Front Surg. 2016 Jan 19;2:71. doi: 10.3389/fsurg.2015.00071. eCollection 2015. PMID 26835456
- [Background] Tzafetta K, Ahmed O, Bahia H, Jerwood D, Ramakrishnan V. Evaluation of the factors related to postmastectomy breast reconstruction. Plast Reconstr Surg. 2001 Jun;107(7):1694-701. doi: 10.1097/00006534-200106000-00009. PMID 11391187
- [Background] Vega S, Smartt JM Jr, Jiang S, Selber JC, Brooks CJM, Herrera HR, Serletti JM. 500 Consecutive patients with free TRAM flap breast reconstruction: a single surgeon's experience. Plast Reconstr Surg. 2008 Aug;122(2):329-339. doi: 10.1097/PRS.0b013e31817f45cb. PMID 18626347
- [Background] Duggal CS, Grudziak J, Metcalfe DB, Carlson GW, Losken A. The effects of breast size in unilateral postmastectomy breast reconstruction. Ann Plast Surg. 2013 May;70(5):506-12. doi: 10.1097/SAP.0b013e318263f1f8. PMID 23542837
- [Background] Noone RB. Thirty-five years of breast reconstruction: eleven lessons to share. Plast Reconstr Surg. 2009 Dec;124(6):1820-1827. doi: 10.1097/PRS.0b013e3181bf821a. No abstract available. PMID 19952638
- [Background] Salzberg CA, Ashikari AY, Koch RM, Chabner-Thompson E. An 8-year experience of direct-to-implant immediate breast reconstruction using human acellular dermal matrix (AlloDerm). Plast Reconstr Surg. 2011 Feb;127(2):514-524. doi: 10.1097/PRS.0b013e318200a961. PMID 21285756
- [Background] Morrison WA, Marre D, Grinsell D, Batty A, Trost N, O'Connor AJ. Creation of a Large Adipose Tissue Construct in Humans Using a Tissue-engineering Chamber: A Step Forward in the Clinical Application of Soft Tissue Engineering. EBioMedicine. 2016 Apr;6:238-245. doi: 10.1016/j.ebiom.2016.03.032. Epub 2016 Mar 23. PMID 27211566
- [Background] Petit JY, Rietjens M, Lohsiriwat V, Rey P, Garusi C, De Lorenzi F, Martella S, Manconi A, Barbieri B, Clough KB. Update on breast reconstruction techniques and indications. World J Surg. 2012 Jul;36(7):1486-97. doi: 10.1007/s00268-012-1486-3. PMID 22395342
- [Background] Cordeiro PG, McCarthy CM. A single surgeon's 12-year experience with tissue expander/implant breast reconstruction: part I. A prospective analysis of early complications. Plast Reconstr Surg. 2006 Sep 15;118(4):825-831. doi: 10.1097/01.prs.0000232362.82402.e8. PMID 16980842
- [Background] Martindale V, Menache A. The PIP scandal: an analysis of the process of quality control that failed to safeguard women from the health risks. J R Soc Med. 2013 May;106(5):173-7. doi: 10.1177/0141076813480994. No abstract available. PMID 23761525
- [Background] Mian R, Morrison WA, Hurley JV, Penington AJ, Romeo R, Tanaka Y, Knight KR. Formation of new tissue from an arteriovenous loop in the absence of added extracellular matrix. Tissue Eng. 2000 Dec;6(6):595-603. doi: 10.1089/10763270050199541. PMID 11103081
- [Background] Tanaka Y, Tsutsumi A, Crowe DM, Tajima S, Morrison WA. Generation of an autologous tissue (matrix) flap by combining an arteriovenous shunt loop with artificial skin in rats: preliminary report. Br J Plast Surg. 2000 Jan;53(1):51-7. doi: 10.1054/bjps.1999.3186. PMID 10657450
- [Background] Hofer SO, Knight KM, Cooper-White JJ, O'Connor AJ, Perera JM, Romeo-Meeuw R, Penington AJ, Knight KR, Morrison WA, Messina A. Increasing the volume of vascularized tissue formation in engineered constructs: an experimental study in rats. Plast Reconstr Surg. 2003 Mar;111(3):1186-92; discussion 1193-4. doi: 10.1097/01.PRS.0000046034.02158.EB. PMID 12621190
- [Background] Cronin KJ, Messina A, Knight KR, Cooper-White JJ, Stevens GW, Penington AJ, Morrison WA. New murine model of spontaneous autologous tissue engineering, combining an arteriovenous pedicle with matrix materials. Plast Reconstr Surg. 2004 Jan;113(1):260-9. doi: 10.1097/01.PRS.0000095942.71618.9D. PMID 14707645
- [Background] Findlay MW, Dolderer JH, Trost N, Craft RO, Cao Y, Cooper-White J, Stevens G, Morrison WA. Tissue-engineered breast reconstruction: bridging the gap toward large-volume tissue engineering in humans. Plast Reconstr Surg. 2011 Dec;128(6):1206-1215. doi: 10.1097/PRS.0b013e318230c5b2. PMID 22094739
- [Background] Findlay MW, Messina A, Thompson EW, Morrison WA. Long-term persistence of tissue-engineered adipose flaps in a murine model to 1 year: an update. Plast Reconstr Surg. 2009 Oct;124(4):1077-1084. doi: 10.1097/PRS.0b013e3181b59ff6. PMID 19935290
- [Background] Faglin P, Gradwohl M, Depoortere C, Germain N, Drucbert AS, Brun S, Nahon C, Dekiouk S, Rech A, Azaroual N, Maboudou P, Payen J, Danze PM, Guerreschi P, Marchetti P. Rationale for the design of 3D-printable bioresorbable tissue-engineering chambers to promote the growth of adipose tissue. Sci Rep. 2020 Jul 16;10(1):11779. doi: 10.1038/s41598-020-68776-8. PMID 32678237
- [Background] Gradwohl M, Chai F, Payen J, Guerreschi P, Marchetti P, Blanchemain N. Effects of Two Melt Extrusion Based Additive Manufacturing Technologies and Common Sterilization Methods on the Properties of a Medical Grade PLGA Copolymer. Polymers (Basel). 2021 Feb 14;13(4):572. doi: 10.3390/polym13040572. PMID 33672918
- [Background] Matsuda K, Falkenberg KJ, Woods AA, Choi YS, Morrison WA, Dilley RJ. Adipose-derived stem cells promote angiogenesis and tissue formation for in vivo tissue engineering. Tissue Eng Part A. 2013 Jun;19(11-12):1327-35. doi: 10.1089/ten.TEA.2012.0391. Epub 2013 Mar 28. PMID 23394225
- See also: Related Info — http://www.who.int/fr/news-room/fact-sheets/detail/breast-cancer